CLINICAL TRIAL: NCT06107634
Title: Can Gastropexy Improve the Efficacy of the Crural Repair in Patients with Paraesophageal Hernias? a Double Blind, Randomized, Multicenter Clinical Trial
Brief Title: Gastropexy in the Repair of Patients with Paraesophageal Hernias
Acronym: PEH3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ersta Diakoni (Other)
Collaborators: Göteborg University (Other); Sundsvall Hospital (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Marcus Reuterwall Hansson, PhD, senior consultant surgeon, Ersta Diakoni
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Dnr 2023-01956-01
Record Dates: First submitted 2023-09-19; First posted 2023-10-30 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Paraesophageal Hernia
MeSH Terms: conditions — Hernia, Hiatal | interventions — Gastropexy

STUDY DESIGN:
Intervention Model Description: Conventional paraesophageal hernia repair with the addition of gastropexy
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization process is initiated after general anesthesia is induced and the group affiliation will be determined by opening of a sealed envelope specifying the group assignment. The information of group allocation is stored in a closed envelope kept in a locked archive until the study is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard paraesophageal hernia repair (Active Comparator): Standard paraesophageal hernia repair (crural suturing and a total (Nissen) fundoplication)
  Interventions: Procedure: Paraesophageal hernia repair
- Standard paraesophageal hernia repair + gastropexy (Experimental): Standard paraesophageal hernia repair with the addition of a three point gastropexy (posterior, left anterolateral and anterior gastropexy)
  Interventions: Procedure: Gastropexy; Procedure: Paraesophageal hernia repair

INTERVENTIONS:
Procedure: Gastropexy — In the intervention group, a three-point gastropexy is added to the repair. First, the right fundus flap is adapted posteriorly to the crural portion of the diaphragm with a 2-3 cm long running non-absorbable suture ("posterior gastropexy"). Second, the left fundus flap is adapted to the diaphragm anterolateral to the hiatus with a 2-3 cm long running non-absorbable suture ("left anterolateral gastropexy"). Finally, the minor curvature of the anterior stomach wall is adapted during reduced intraabdominal pressure to the anterior abdominal wall with a 2-3 cm long running non-absorbable suture ("anterior gastropexy").
  Arms: Standard paraesophageal hernia repair + gastropexy
Procedure: Paraesophageal hernia repair — Ultrasonic shears are used for dissection. The herniated viscera are completely reduced into the abdomen and the hernia sac in fully dissected and resected. The esophagus is mobilized intraabdominally until at least 3 cm rests below the hiatus without tension. The anterior and posterior vagal nerves are identified and preserved. A posterior crural closure with running non-absorbable sutures is performed. An additional anterior crural closure may be performed at the surgeon's discretion. The fundus is mobilized to allow a floppy fundoplication. A total fundoplication is created by three interrupted non-absorbable sutures. No bougies are used routinely for calibration of the fundoplication.

SUMMARY:
Patients scheduled for surgery for primary paraesophageal herniation are randomized to either conventional surgical hernia repair or with the addition of gastropexy.

DETAILED DESCRIPTION:
Patients scheduled for surgery due to primary paraesophageal herniation are randomized into either the control group or the interventional group.

Control Group: Patients undergo a crural repair combined with a short and floppy Nissen fundoplication.

Interventional Group: In addition to the crural repair and Nissen fundoplication, patients receive a gastropexy. This involves the fixation of the posterior part of the wrap the right crus, the left portion of the wrap to the diaphragm, and the minor curvature of the stomach to the abdominal wall.

Follow-Up Assessments:

Imaging: Computed tomography (CT) scans are performed before surgery and at 1 and 3 years postoperatively to evaluate anatomical outcomes.

Patient-Reported Outcomes: The following questionnaires are completed before surgery, as well as at 3 months, 1 year, and 3 years after surgery:

SF-36: A global quality of life instrument. GSRS: The Gastrointestinal Symptoms Rating Scale. Reflux Frequency Questionnaire: A measure reflux disease-related symptoms. Dakkak's Dysphagia Score: An assessment of swallowing difficulties.

ELIGIBILITY:
Inclusion Criteria:

- Patients diagnosed with a primary paraesophageal hernia (hiatal hernia types II-IV) who are scheduled for elective or emergency surgical repair at participating centers

Exclusion Criteria:

* Previous major upper gastrointestinal (GI) surgery, including prior hiatal hernia repair.
* Diagnosis of achalasia or any other significant esophageal motility disorder.
* Inability to understand the purpose of the study and/or inability or unwillingness to provide informed consent.
* Severe comorbidities, defined by an American Society of Anesthesiologists (ASA) physical status score of greater than III.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-08-02 (Estimated); Study Completion 2030-08-02 (Estimated)

PRIMARY OUTCOMES:
Recurrence of hernia at 1 year after surgery | 1 year
  Computer tomography of abdomen and thorax

SECONDARY OUTCOMES:
Recurrence of hernia at 3 years after surgery | 3 year
  Computer tomography of abdomen and thorax
Complications after surgery | 30 days after surgery
  Complication classified according to Clavien-Dindo
Length of stay at the hospital after surgery | 30 days after surgery
  Information from patients journal
Changes in the patients perception of quality of life after surgery | 3 months, 12 months, and 36 months
  SF-36 (Short Form 36) is a health related quality of life questionnaire. SF-36 is comprised of 36 items that assess eight dimensions of health: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions. Higher scores mean a better outcome. These can be grouped into mental and physical component summary scores. Scoring is from 0-100. A mean score of 50 has been articulated as normative value.
Changes in the patients perception of gastrointestinal symptoms after surgery | 3 months, 12 months, and 36 months
  GSRS (The Gastrointestinal Symptom Rating Scale) is a questionnaire, which contains 15 items, and uses a seven-graded Likert scale, where 1 represents the most positive option and 7 the most negative one. The questions are grouped in five dimensions. A mean value for the items in each dimension will be calculated:
  Diarrhoea syndrome: 11. Increased passage of stools 12. Loose stools 14. Urgent need for defecation
  Indigestion syndrome: 6. Borborygmus 7. Abdominal distension 8. Eructation 9. Increased flatus
  Constipation syndrome: 10. Decreased passage of stools 13. Hard stools 15. Feeling of incomplete evacuation
  Abdominal pain syndrome: 1. Abdominal pain 4. Sucking sensations 5. Nausea and vomiting
  Reflux syndrome: 2. Heartburn 3. Acid regurgitation.
Changes in the patients perception of dysphagia after surgery | 3 months, 12 months, and 36 months
  The Dakkak dysphagia score is a questionnaire for assessing benign dysphagia, including nine questions regarding the frequency (always, sometimes, or never) of swallowing difficulties with different food consistencies (liquid, semisolid, and solid foods). The final score ranges from 0 to 45, where 45 represents the most severe dysphagia.
Changes in the patients perception of dysphagia and reflux frequency after surgery | 3 months, 12 months, and 36 months
  Symptoms of heartburn, reflux, chest pain, dysphagia for liquids and solids, dyspnea, coughing and odynophagia were recorded using a four-graded scale to assess the frequency of symptoms with an arbitrary (empirical) cut off for clinical significance. The same instrument has been used in a previous RCT, from the same institution, comparing different types of anti-reflux procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Thorell, Professor, Study Director — Ersta Diakoni
Locations (6):
- Sweden (6):
  - Sahlgrenska University Hospital, Gothenburg
  - Skåne University Hospital Lund, Lund
  - Nyköping Hospital, Nyköping
  - Ersta Hospital, Stockholm
  - Sundsvall County Hospital, Sundsvall
  - Uppsala Academic Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No